CLINICAL TRIAL: NCT06560359
Title: Neurobehavioral Effects of Increased Fruit and Vegetable Intake on Cognition, Mood, and Attention in 7-11-Year-Old Children From Shanghai: A Randomized Controlled Trial
Brief Title: RCT on the Neurobehavioral Effects of Fruits and Vegetables in Shanghai Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Chen, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HN25462
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Function; Mood Disorders; Attention-deficit
MeSH Terms: conditions — Mood Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Two groups (Trial group and Control group) start with 2 weeks of no F&V, following 12 weeks of intervention, and then 4-6 weeks of washout (both groups with no intervention), this full study takes 18 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trial Group (Experimental): Participants in the Trial Group will receive a daily intervention consisting of a breakfast that includes one piece of fruits (e.g., an apple or a banana), vegetables (e.g., a carrot or a cucumber), and other regular diet. The fruit and vegetable will be provided as part of a standardized breakfast menu designed by nutrition experts. This intervention will be administered every morning, seven days a week, for a duration of 12 weeks. The goal is to increase the daily intake of fruits and vegetables among participants to assess the effects on cognitive performance, mood and attention.
  Interventions: Dietary Supplement: F&V
- Control group (Placebo Comparator): Participants in the Control Group will maintain their regular breakfast without any additional interventions related to fruit and vegetable intake. No changes will be made to their daily breakfast routine.
  Interventions: Dietary Supplement: No F&V

INTERVENTIONS:
Dietary Supplement: F&V — The intervention includes the healthy breakfast plan (daily delivery of balanced breakfast containing at least one piece of fruits, vegetables and other regular diet). Meals were centrally prepared by a professional catering service and delivered every morning, seven days a week, to participants' homes, ensuring consistency in portion size and quality. The selection of fruits and vegetables will consider seasonal availability to ensure freshness and variety. Nutrient density and adequacy will be monitored throughout the intervention period, with adjustments made as needed to maintain the nutritional integrity of the meals. Compliance will be tracked through daily logs and periodic assessments, ensuring that participants are consistently consuming the provided meals. This intervention is specifically designed to investigate the neurobehavioral impact of increased fruit and vegetable intake in a controlled and measurable manner.
  Arms: Trial Group
Dietary Supplement: No F&V — The intervention only includes breakfast plan (daily delivery of balanced breakfast containing regular diet without fruits and vegetables) for 12 weeks. Meals were centrally prepared by a professional catering service and delivered every morning, seven days a week, to participants' homes, ensuring consistency in portion size and quality. Nutrient density and adequacy will be monitored throughout the intervention period, with adjustments made as needed to maintain the nutritional integrity of the meals. Compliance will be tracked through daily logs and periodic assessments, ensuring that participants are consistently consuming the provided meals. This intervention is specifically designed to investigate the neurobehavioral impact of increased fruit and vegetable intake in a controlled and measurable manner.
  Arms: Control group

SUMMARY:
This project proposal outlines a randomized-controlled trial (RCT) aimed at evaluating the effects of increased fruit and vegetable (F&V) intake on cognitive performance, attention, and mood in Chinese children aged 7-11 years. The increased F&V intake will be achieved by providing a daily healthy breakfast including at least one piece of fruits and one piece of vegetables. The RCT includes a 2-week Lead-In term, 12 week Intervention term and 4-6 week Washout/Follow-Up term, targeting 250 children from the selected schools in Shanghai. The primary objective is to measure cognitive improvement using the Wechsler Intelligence Scale for Children (WISC-IV), while secondary outcomes will assess mood, attention, biomarkers, behavioral changes in dietary choices and the mechanism. The results of this trial may provide critical evidence on the benefits of F&V consumption in children.

DETAILED DESCRIPTION:
1. Intervention Method: The intervention will be implemented through the Healthy Breakfast Plan.

   1. Healthy Breakfast Plan: During the 12-week intervention period, a pre-designed breakfast (including regular breakfast foods with fruits and vegetables) will be delivered daily to the homes of participating children.
   2. Important Considerations:

   i) The Breakfast Plan will include both the intervention group and the control group. The intervention group will receive the intervention meal (having fruits and vegetables), while the control group will receive a control meal (not having fruits and vegetables).

   ii) The nutritional composition of the Healthy Breakfast Plan will be pre-designed by experts from the Department of Nutrition and Food Hygiene at Fudan University to ensure scientific accuracy.
2. Sample Size: The study will include a total of 250 children from the selected schools. Children will be randomly selected from 6 to 8 classes, resulting in approximately 125 children in the trial group and 125 in the control group. Cluster randomization will be applied at the classroom level, ensuring that all children within the same classroom are assigned to the same group. The sample size calculation is based on previous studies of literature using the Wechsler Intelligence Scale for Children (WISC-IV) to assess cognitive function. With assumptions based on existing literature, the study requires at least 150 participants to achieve statistical power. Accounting for a 20% attrition rate, a sample size of 188 is chosen to ensure robustness.
3. Exposure: Biomarkers, specifically vitamin C (ascorbic acid), will be measured from urine samples to monitor the intake of fruits and vegetables. The analysis will be conducted using reverse-phase high-performance liquid chromatography (HPLC) with UV detection or ultra-performance liquid chromatography coupled with mass spectrometry (UPLC-MS/MS).
4. Quality Control: To ensure accuracy in dietary intake reporting, the study will utilize food frequency questionnaires and 24-hour dietary records. These tools will help monitor and validate the children's fruit and vegetable consumption throughout the intervention period.
5. Ensuring Compliance with Fruit and Vegetable Intake:

   1. Vitamin C Measurement: Urinary vitamin C levels will be measured to verify actual fruit and vegetable intake.
   2. Questionnaires: Supervision of intake will be supported by questionnaires designed to track compliance and dietary habits.
   3. Online Management Software: The study will use online management software to document each aspect of the project, allowing the research team and supervisors to monitor progress in real-time.
6. Data Collection and Assessments:

   (a) Survey Questionnaires: i) Cognition: Evaluated by Wechsler Intelligence Scale for Children (WISC-IV). ii) Mood: Evaluated using the Profile of Mood States (POMS) questionnaire. iii) Attention: Evaluated by the Conners Parent Symptom Questionnaire (PSQ). iv) Physical Activity: Assessed using the International Physical Activity Questionnaire (IPAQ).

   v) Dietary Habits and Preferences: Assessed by Food Frequency Questionnaire (FFQ), 24-hour dietary records, and the food preference questionnaires.

   (b) Biological Specimen Collection: i) Urine sample: for measuring vitamin C. ii) Saliva sample: for measuring cortisol. Saliva sample will be collected from a subpopulation as a pilot study.

   iii) Feces: for exploring the gut mechanisms that may modify the neurobehavior effects by increased intake of fruits and vegetables. Feces sample will be collected from a subpopulation as a pilot study.

   (c) Physical Examinations: i) Measurements of height, weight, waist-to-hip ratio, and skinfold thickness will be taken to assess the overall physical health of participants.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-11 years.
* Participants must be students enrolled in the selected schools participating in the study.
* Willingness and ability to consume the provided daily breakfast, including one piece of fruit and one piece of vegetable.
* Parents or legal guardians must provide informed consent for participation.
* Balanced preliminary investigation outcomes, especially regarding behaviors related to fruit and vegetable intake, socioeconomic status (SES), and absence of diagnosed diseases that could impact the study.

Exclusion Criteria:

* Known allergies to any fruits, vegetables, or other foods provided in the intervention.
* Diagnosed psychological disorders, diabetes, gastrointestinal diseases, or other conditions that might interfere with cognitive assessments or the ability to participate in the study.
* Children currently participating in other dietary or cognitive intervention studies.
* Inability or unwillingness to comply with study protocols, including dietary requirements and sample collection.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Performance | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  The primary outcome measure will assess the change in cognitive performance of children participating in the study. This will be evaluated using the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV), which is validated for use with Chinese children. The WISC-IV scale includes a range of cognitive tests that produce a Full Scale IQ score, with subtests for Verbal Comprehension, Perceptual Reasoning, Working Memory, and Processing Speed. The scores range from 40 to 160, where higher scores indicate better cognitive performance. The measure will focus on the change in cognitive scores from baseline to post-intervention, as well as the retention of any cognitive changes after the washout period.

SECONDARY OUTCOMES:
Change in Mood States | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  This outcome will measure the change in mood states among participants, using the Profile of Mood States (POMS) questionnaire, which is validated for use in Chinese children. The POMS questionnaire assesses various aspects of mood, including tension, depression, anger, vigor, fatigue, and confusion. The scores for each mood state range from 0 to 4, with higher scores indicating a worse outcome in negative mood states (tension, depression, anger, fatigue, and confusion) and a better outcome in the positive mood state (vigor).
Change in Attention | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  This outcome will assess changes in attention among participants, as perceived by their parents, using the Conners' Parent Rating Scale (CPRS), which is also referred to in some contexts as the Conners Parent Symptom Questionnaire (PSQ). The CPRS is a validated tool used in the Chinese population to evaluate behavioral concerns, including attention. The scale includes items rated on a 4-point Likert scale, with scores ranging from 0 (Not at all true) to 3 (Very much true). Higher scores indicating worse attention outcomes, i.e., more attention-related problems.
Identification of Biomarkers in Saliva, Urine, and Feces Related to Cognition, Mood, and Attention | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  Vitamin C in urine will be served as a biomarker of F&V intake. The biomarkers in saliva and feces will be served as the indicators of cognitive function, mood states, or attention levels. Samples of saliva and feces will be collected in a subpopulation as a pilot study. These biomarkers will be analyzed to understand the physiological changes associated with increased fruit and vegetable intake.
Behavioral Changes in Dietary Choices Influenced by Fruit and Vegetable Intake | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  This outcome will evaluate how increased intake of fruits and vegetables impacts dietary behavior, specifically the choices participants make regarding their overall diet. The assessment will be conducted using validated questionnaires that capture changes in dietary habits and preferences.
Investigation of Current Status and Barriers to Fruit and Vegetable Intake | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  This objective aims to assess the current level of fruit and vegetable intake among children and identify the barriers that limit their consumption. Factors such as nutrition literacy, food accessibility, and socioeconomic status will be explored to understand the challenges and opportunities for improving F&V intake in this population.
Mechanistic Study of Cognitive Effects through Gut Microbiota | the end of Week 2 (Baseline), Week 14 (end of intervention), and Week 18-20 (post-washout).
  This outcome will only be measured in a subpopulation as a pilot study, which will will investigate the mechanisms by which increased fruit and vegetable intake influences cognitive function. The study will assess changes in gut microbiota composition through stool samples.

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No